CLINICAL TRIAL: NCT02855736
Title: Effectiveness of Positive Psychology in Suicidal Patients: A Randomized Controlled Trial
Brief Title: Positive Psychology in Suicidal Patients
Acronym: POPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UF 9557; 2015-A00358-41 (Other: FRANCE: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-07-08; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Suicidal Thoughts; Suicidal Crisis
Keywords: Suicidal inpatients; Positive Psychology; Gratitude; Psychological pain
MeSH Terms: conditions — Suicidal Ideation | interventions — Psychology, Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Positive Psychology (gratitude journal)
  Interventions: Behavioral: Positive Psychology
- Control group (Placebo Comparator): Alimentary list
  Interventions: Behavioral: Placebo (food journal)

INTERVENTIONS:
Behavioral: Positive Psychology — Gratitude Journal (Emmons and Stern, 2013)
  Every evening, patients have to write down the things they feel grateful about.
  Arms: Intervention group
Behavioral: Placebo (food journal) — Food journal (i.e. alimentary list):
  Patients have to write down the list of foods eaten during the day.
  Arms: Control group

SUMMARY:
Suicide is a major health concern. Weeks following psychiatric admission are a highly suicide risk period for those having current suicidal ideation or attempt. Recently, a pilot study suggested the feasibility of positive psychology in patients in suicidal crisis. Notably, gratitude exercises suggested improvement in optimism and hopelessness, two dimensions associated to suicide. Moreover, gratitude has been associated to suicidal ideation and attempt, independently from depression. Thus, investigators want to conduct the first randomized controlled study in order to assess effectiveness of gratitude exercises (vs control task) in suicidal inpatients, on 1) psychological pain reduction 2) suicidal ideation, hopelessness, optimism, depressive symptomatology, and anxiety improvement.

DETAILED DESCRIPTION:
Study design: monocentric randomized controlled study

Methods:

206 inpatients (Department of Emergency Psychiatry and Post Acute Care), between 18 and 65 years-old, having attempted suicide before hospitalisation or having current active suicidal ideation at the time of the psychiatric hospitalisation. Patients suffering from schizophrenia are excluded.

Randomization into two groups: Positive Psychology (i.e., gratitude journal) (n = 103) or Control Task (i.e., food journal) (n = 103), daily exercises during 7 days (in add-on from usual treatment).

Clinical assessment: 1) at baseline (the day before the intervention beginning) (V0); 2) short daily self-assessments (immediately before and after the exercise); 3) the day following the last day of the intervention (V1).

* V0 : socio-demographic data, treatments, psychopathology, suicidal ideation,depressive and anxious symptomatology, psychological pain, optimism, hopelessness.
* Daily self-assessments: psychological pain, optimism, hopelessness
* V1 : treatments suicidal ideation,depressive and anxious symptomatology, psychological pain, optimism, hopelessness, intervention satisfaction.

ELIGIBILITY:
Inclusion criteria:

* Being hospitalized for suicidal thoughts or suicide attempt (from less than a week)
* Having signed informed consent
* Be fluent in French
* Able to understand nature, aims and methodology of the study

Exclusion criteria:

* Lifetime history of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders - V (DSM-V) criteria
* Current eating disorder according to DSM-V criteria
* Patient on protective measures (guardianship or trusteeship)
* Deprived of liberty subject (judicial or administrative decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Psychological pain reduction using a likert scale | At the inclusion and day 8 (the day after the end of the intervention)
  Psychological pain reduction, in gratitude vs control group, between the beginning and the end of the intervention, using a likert scale.

SECONDARY OUTCOMES:
Psychological pain reduction using a likert scale | At day 1, 2, 3, 4, 5, 6, 7
  Psychological pain reduction, in gratitude vs control group, the beginning and the end of each exercise, using a likert scale.
intensity of suicidal ideation | At the inclusion and day 8 (the day after the end of the intervention)
  Reduction of suicidal ideation intensity, in gratitude vs control group between the beginning and the end of the intervention using a Likert Scale and the Scale for Suicidal Ideation (SSI).
Intensity of hopelessness | At the inclusion and day 8 (the day after the end of the intervention)
  Reduction of hopelessness, in gratitude vs control group between the beginning and the end of the intervention, using a Likert Scale and the Beck Hopelessness Scale (BHS).
Intensity of optimism | At the inclusion and day 8 (the day after the end of the intervention)
  Reduction of hopelessness, in gratitude vs control group between the beginning and the end of the intervention, using a Likert Scale and the Life Orientation Test-Revised (LOT-R).
Intensity of depressive symptoms using the Beck Depression Inventory (BDI) | Day 8 (the day after the end of the intervention)
  Reduction of depressive symptoms between the beginning and the end of the intervention, using the Beck Depression Inventory (BDI)
Intensity of anxious symptoms using the State Anxiety Inventory- State (SAI-State) | Day 8 (the day after the end of the intervention)
  Reduction of anxious symptoms between the beginning and the end of the intervention, using the State Anxiety Inventory- State (SAI-State)
Perceived usefulness of the intervention using a likert scale | Day 8 (the day after the end of the intervention)
  Evaluation of the perceived usefulness of each intervention, using a likert scale.
Intensity of suicidal ideation | At day 1, 2, 3,4 5, 6, 7
  Reduction of suicidal ideation intensity, in gratitude vs control group between the beginning and the end of each exercise, using a Likert Scale.
Intensity of hopelessness | At day 1, 2, 3, 4, 5, 6, 7
  Reduction of hopelessness, in gratitude vs control group between the beginning and the end of each exercise, using a Likert Scale.
Intensity of optimism | At day 1, 2, 3, 4, 5, 6, 7
  Reduction of hopelessness, in gratitude vs control group between the beginning and the end of each exercise, using a Likert Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No